CLINICAL TRIAL: NCT00098527
Title: A Phase 2 Study of Single Agent Depsipeptide (FK228) in Gastric and Esophageal Cancers
Brief Title: FR901228 in Treating Patients With Refractory Stomach Cancer or Gastroesophageal Junction Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02637; 6075-04-7R0; DUMC-6075-04-7R0; CDR0000398177; NCI-6351; U01CA099118 (NIH)
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Adenocarcinoma of the Esophagus; Adenocarcinoma of the Stomach; Recurrent Esophageal Cancer; Recurrent Gastric Cancer
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Neoplasms; Stomach Neoplasms | interventions — romidepsin

ARMS (1):
- Treatment (romidepsin) (Experimental): Patients receive FR901228 (depsipeptide) IV over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: romidepsin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: romidepsin — Given IV
  Other Names: FK228; FR901228; Istodax
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well FR901228 works in treating patients with refractory stomach cancer or gastroesophageal junction. Drugs used in chemotherapy, such as FR901228, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. FR901228 may also stop the growth of tumor cells by blocking some of the enzymes needed for their growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the radiographic response rate (complete response and partial response) in patients with refractory adenocarcinoma of the stomach or gastroesophageal junction treated with FR901228 (depsipeptide).

SECONDARY OBJECTIVES:

I. Determine the median time to progression and progression-free survival of patients treated with this drug.

II. Determine the grade 3 and 4 toxic effects of this drug in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive FR901228 (depsipeptide) IV over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 13-20 patients will be accrued for this study within 6.5-10 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the stomach or gastroesophageal junction
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* Refractory* to at least 1, but no more than 3, of the following first-line agents:

  * Fluoropyrimidine (e.g., capecitabine or fluorouracil)
  * Taxane (e.g., paclitaxel or docetaxel)
  * Platinum (e.g., carboplatin, cisplatin, or oxaliplatin)
* No known active brain metastases

  * Treated brain metastases allowed provided metastases are stable off steroids for ≥ 30 days
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* At least 3 months
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN (5 times ULN if liver metastases are present)
* Creatinine clearance ≥ 50 mL/min
* No congestive heart failure
* No New York Heart Association class III or IV heart disease
* No myocardial infarction within the past 6 months
* No ventricular arrhythmias requiring medication
* No angioplasty or vascular stenting within the past 3 months
* No unstable angina
* No left ventricular hypertrophy by EKG
* No known history of serious ventricular arrhythmia (e.g., ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row)
* QTc < 500 msec
* LVEF > 40% by MUGA or echocardiogram
* No other significant cardiac disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Potassium ≥ 4.0 mmol/L (stable level with no change in supplementation within the past 2 weeks)
* Magnesium ≥ 2.0 mg/dL (stable level with no change in supplementation within the past 2 weeks)
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to study drug
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* Prior biological agents allowed
* No concurrent prophylactic filgrastim (G-CSF)
* No concurrent biologic therapy
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No other concurrent chemotherapy
* More than 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy
* Prior targeted agents allowed
* No other prior or concurrent cytotoxic agents
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No concurrent medications causing QTc prolongation
* No concurrent potassium supplementation > 40 mg/day or magnesium supplementation > 1 g/week
* No concurrent hydrochlorothiazide
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-10; Primary Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Radiographic response rate (complete response & partial response) | Not Provided

SECONDARY OUTCOMES:
Progression-free survival (PFS) according to RECIST | Up to more than 6 months
  The median time to progression and median PFS for all eligible patients, along with their CIs, will be reported. The Kaplan-Meier analysis approach may be used to summarize these time-to-event endpoints.
Frequency of treatment related grade 1-4 toxicities and cardiac toxicities as assessed by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | Up to 12 months
Correlation of changes in gene expression profile in dermal granulation tissue pre- and post-treatment with gene expression profile | Not Provided
Correlation of wound vascular scores pre- and post-treatment with gene/protein changes | Not Provided
Toxicity | Not Provided
Changes in gene expression profile | At pre- and post-treatment
Changes in levels of p21 and thymidine kinase expression, and tubulin acetylation using Western blotting | From baseline to 3 weeks
Changes in gene expression profile in dermal granulation tissue | From baseline to up to 3 weeks
Change in plasma and urine TGFB levels | At pre-and post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Hurwitz, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States